CLINICAL TRIAL: NCT07224620
Title: Fentanyl Versus Hydromorphone as First Line Strategy in Patients on Mechanical Ventilation, a Pilot Pragmatic Randomized Superiority Clinical Trial: the FenHydro Trial
Brief Title: Fentanyl Versus Hydromorphone in Patients on Mechanical Ventilation
Acronym: FenHydro
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Elias Baedorf Kassis, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P000456
Record Dates: First submitted 2025-10-28; First posted 2025-11-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Mechanical Ventilation; Sedation and Analgesia; Critical Care, Intensive Care
Keywords: Fentanyl; Hydromorphone; Mechanical ventilation; Intensive Care Unit; ICU; Analgosedation; Analgesia; Sedation
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Hydromorphone

STUDY DESIGN:
Intervention Model Description: Randomization will occur at the level of the ICU, rather than for each individual patient. Cluster I (MICU A, B, C) and cluster II (FICU) will be randomized to start from a period with fentanyl or hydromorphone and after 3 months will be crossed over to the other group. The process will be repeated during the study period. Cluster cross-over are planned to be 3 months to avoid seasonal variability. The investigators plan to start the enrollment in the middle of a season, so that the clusters have 1.5 months of each season. No washout period is planned.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl as first line agent (Experimental): Patients in an ICU on a three-month period randomized to Fentanyl will have Fentanyl used as suggested first-line therapy for analgosedation, when clinically warranted.
  Interventions: Drug: fentanyl
- Hydromorphone as first line agent (Experimental): Patients in an ICU on a three-month period randomized to Hydromorphone will have Hydromorphone used as suggested first-line therapy for analgosedation, when clinically warranted.
  Interventions: Drug: Hydromorphone

INTERVENTIONS:
Drug: fentanyl — Suggested initial continuous infusion
  * Route: Intravenous
  * Dose: 0-200 mcg/hr (max 1,440 MME/day)
  * Initial dose: 50mcg/hr
  * Concentration: 50 mcg/mL
  * Bolus: 50-200mcg up to every 5 minutes as needed
  * Continuous infusion adjustment: Increase in the continuous infusion if sedation not at goal after 3 bolus doses, increase by 25 mcg/hr every 60 minutes
  Titration of dose, initial dose, adjustments and bolus are just suggested. The primary team is allowed to modify them based on clinical judgement.
  Arms: Fentanyl as first line agent
Drug: Hydromorphone — Suggested initial continuous infusion
  * Route: Intravenous
  * Dose: 0-3 mg/hr (max 1,440 MME/day)
  * Initial dose: 0.5mg/hr
  * Concentration: 0.2 mg/mL
  * Bolus: 0.5-2mg up to every 5 minutes as needed
  * Continuous infusion adjustment: Increase in the continuous infusion if sedation not at goal after 3 bolus doses, increase by 0.25 mg/hr every 60 minutes
  Titration of dose, initial dose, adjustments and bolus are just suggested. The primary team is allowed to modify them based on clinical judgement.
  Other Names: Dilaudid
  Arms: Hydromorphone as first line agent

SUMMARY:
Patients with respiratory failure who require mechanical ventilation are not only at risk of death, but also of complications of prolonged ICU stay. Patients may have significant functional decline, impact in quality of life, develop psychiatric disorders and at long-term can lead to significant cost to society. Although sedation and analgesia are considered only supportive therapy, several studies have shown that in patients on mechanical ventilation, different approaches can have significant impact on patient centered outcomes. However, to date, randomized clinical trials on critically ill patients have mostly evaluated the sedative agent but not the analgesic agent. Although morphine and its derivates are the most common used opioid analgesic agents in the critical care setting, only some retrospective studies and some prospective studies compared them head-to-head (ramifentanyl versus morphine and fentanyl versus morphine). Current guidelines recommend choosing the analgesic agent based on pharmacokinectics, physician experience and side-effects profile. To evaluate the differences of two standard-of-care analgosedation agents, the FenHydro trial will be a cluster randomized, pragmatic, pilot and feasibility superiority clinical trial in mechanically ventilated patients in the ICU. The main question the study hopes to answer is whether there is any difference in morphine milligram equivalents administered during mechanical ventilation.

DETAILED DESCRIPTION:
Fentanyl is a synthetic derivate of morphine that is 100 times more potent than morphine, has a great lipid solubility leading to fast onset (one to two minutes), has a short half-life (up to three hours) and limited histamine release. It is metabolized by the liver and its excretion is not affected by the kidneys. Those characteristics allow fentanyl to be versatile and be used in many different scenarios in the ICU. Despite those advantages, concerns have been raised regarding adipose tissue accumulation, tachyphylaxis, CYP3A4 interaction and chest wall rigidity, particularly when on high doses.

Hydromorphone is an alternative analgesic agent. It is a semisynthetic morphine derivate that can be five to ten times more potent than morphine. It also has a fast onset (up to 10 minutes), a short half-life (up to three hours) and is less renally excreted than morphine. Some concerns have been raised regarding the accumulation of hydromorphone metabolites including hydromorphone-3-glucuronide, which can lead to neuroexcitatory effects and delirium. A few retrospective studies compared fentanyl and hydromorphone in the critical care setting. Due to the retrospective nature, small size of the studies and several imbalances in the groups, no significant conclusion can be drawn regarding the benefits and risks of fentanyl versus hydromorphone. However, the largest and most recent retrospective study, showed no difference in 28-day mechanical ventilation free days and death during mechanical ventilation.

Opioids currently used for analgosedation in mechanically ventilated ICU patients include morphine, fentanyl and hydromorphone. The selection of a specific agent as standard-of-care is determined by primary ICU team preference, logistics, patient characteristics and experience. Although small differences may affect the decision of one over the other, dosage reduction and close monitoring are used rather than switching to an alternative in most cases. Whether or not either of these agents afford additional meaningful clinical benefits, advantages or contribute to meaningful clinical outcomes has not been fully established in available literature and represents the basis for performing this clinical pilot study. Therefore, the investigators propose to study the use of fentanyl and hydromorphone in the critically ill population on mechanical ventilation due to the paucity of data comparing both medications head-to-head and their widespread use.

Between November 2025 and April 2026, all patients on mechanical ventilation admitted to the medical intensive care units (MICU) and Finard intensive care unit (FICU - medical and surgical ICU) at Beth Israel Deaconess Medical Center who are 18 years or older will be enrolled. The study will be pragmatic and randomization will be in two clusters. The MICU and the FICU will be randomized to an initial opioid (fentanyl or hydromorphone) in three-months blocks. The assigned opioid will be used as the first line agent of choice for analgosedation. The assigned opioid will be switched at the end of the three-months block. Since the study has a 6 months duration, each ICU will have 3 months with each opioid as first line for analgosedation. The investigators anticipate that 300 patients will be required for sample size.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to either MICU A, B, C or FICU at Beth Israel Deaconess Medical Center
* Requiring mechanical ventilation
* Felt by primary team to require opioid infusion for analgosedation

Exclusion Criteria:

* Age < 18 years old
* Do not intubate orders prior to enrollment
* Comfort measures only
* Contraindication to fentanyl or hydromorphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Difference in daily MME dose received during mechanical ventilation period. | Assessed from enrollment (baseline) censored at day 28
  The daily MME dose will be calculated using all the opioid doses received during the day. The outcome will be obtained from the days patients were on mechanical ventilation. It will include not only the intervention medication, but also the additional boluses and alternate opioids, including cross-over drug. The doses will be converted into MME.

SECONDARY OUTCOMES:
All cause 28-day hospital mortality | 28 days after enrollment censored at hospital discharge
  Death before hospital discharge. Patients who were discharged prior to 28 days will be assumed to be alive.
Days alive and free of mechanical ventilation at day 28 | 28 days after enrollment censored at hospital discharge
  The ventilator free days will be counted as 28 minus the duration of mechanical ventilation in days for those patients who survived the 28 days. Patients discharged prior to 28 days will be assumed to be free of mechanical ventilation. Patients who died before 28 days will be assumed to have zero ventilation free days
Days alive and free of ICU at day 28 | 28 days after enrollment censored at hospital discharge
  Counted as 28 minus the days alive in the ICU. Patients discharged prior to 28 days will be assumed to be out of the ICU. Patients who died before 28 days will be assumed as zero ICU free days
Days alive and free of vasopressors at day 28 | 28 days after enrollment censored at hospital discharge
  Counted as 28 minus the days alive with intravenous vasopressors. Patients discharged prior to 28 days will be assumed to be off of vasopressors. Patients who die before 28 days will be assumed as zero vasopressors free days
Difference in average daily dose of morphine milligram equivalent required during the first 28 days | 28 days after enrollment censored at hospital discharge
  Will be calculated based on daily average dose through 28 days of the intervention drug and other opioids received during hospital admission. The dose of opioids used on the comfort measures period for those patients that were transitioned to comfort measures will not be considered for the outcome analysis. Patients discharged prior to 28 days of enrollment will be considered to have 0 morphine milligram equivalent per day after discharge.
Percentage of time without coma and delirium during the ICU stay | Assessed from enrollment (baseline) censored at day 28
  Assessed daily by RASS and CAM-ICU by nurses at the bedside during ICU stay. A positive day for coma is RASS of -3 or less and delirium is considered as RASS of 3 or more or positive CAM-ICU. Percentage will be obtained by dividing the number of days without coma and delirium by the numbers of ICU days.
Days alive and free of restraints at 28 days | 28 days after enrollment censored at hospital discharge
  Counted as 28 minus the days alive with need for restraints. Patients discharged prior to 28 days will be assumed to be off of restraints. Patients who die before 28 days will be assumed as zero restraints free days.
Daily Average number of Bowel Movements through ICU stay | Assessed from enrollment (baseline) censored at day 28
  Will be measured by the number of bowel movements per day during the ICU stay. In patients with rectal tube, 1 bowel movement will be considered to have least 100mL and a maximum of 250mL of stools.
Need for tracheostomy during hospital stay or 28 days | Hospital stay or 28 days (whichever comes first)
  Incidence of tracheostomy required during hospital stay or 28 days
Days alive and out of hospital | 28 days after enrollment censored at hospital discharge
  Counted as 28 minus the days alive in the hospital. Patients who died before 28 days will be assumed as zero ICU free days

OTHER OUTCOMES:
Requirement of adjunctive analgesia or sedation medications | Measured through 28 days after enrollment.
  Total dose and medications used during 28 days in propofol equivalent dose. Patients discharged before the day 28th will be considered to be on no sedative medication.
Patient-ventilator respiratory mechanics | Through mechanical ventilation period in the first 3 and 7 days
  The investigators will measure and compare respiratory mechanics. They will be measured daily during the MV period, per primary team decision. The investigators will compare the weighted average of PEEP, plateau, compliance and driving pressure during in the first 3 days and in the first 7 days.
Mean difference in total MME dose received during the first 24 hours, first 3 days | Day 1, 3 and 7 after enrollment
  Will be calculated based on total dose at day 1, 3 and 7 after enrollment. Will include all opioids used in MME. The dose of opioids used on the comfort measures period for those patients that were transitioned to comfort measures will not be considered for the outcome analysis. Patients discharged prior to day 1, 3 or 7 after enrollment will be considered to have 0 MME per day.
Mean Daily Vasopressor Dose | Assessed from enrollment (baseline) censored at day 28
  Difference in mean Daily Vasopressor dose in norepinephrine equivalents measured during ICU stay. The daily vasopressor dose will be calculated using all the vasopressors received during the day (eg, norepinephrine, vasopressin, dobutamine, epinephrine, phenylephrine, angiotensin II).

CONTACTS AND LOCATIONS:
Overall Officials: Elias N Baedorf-Kassis, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for secondary use of the dataset can be made by emailing Dr. Eduardo Padrao. The data available will be identified.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Individual participant data that underlie the results will be available starting 12 months after publication of the main results paper and will remain available for 5 years after that date
Access Criteria: Who can access the data: Data will be made available to researchers whose proposed use of the data has been approved by the lead trial investigators.
  Types of analyses: For any purpose that facilitates advancement of the field Mechanisms of data availability: With investigator support and IRB approval, after approval of a proposal, with a signed data access agreement